CLINICAL TRIAL: NCT03341143
Title: Phase II Feasibility Study of Fecal Microbiota Transplant (FMT) in Advanced Melanoma Patients Not Responding to PD-1 Blockade
Brief Title: Fecal Microbiota Transplant (FMT) in Melanoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zarour, Hassane, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Diwakar Davar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 17-034
Record Dates: First submitted 2017-09-28; First posted 2017-11-14 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Melanoma
Keywords: Unresectable; Stage III; Stage IV
MeSH Terms: conditions — Melanoma | interventions — Fecal Microbiota Transplantation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fecal Microbiota Transplant (FMT) with Pembrolizumab (Experimental): The FMT along with an intestinal biopsy will be performed as outpatient by a gastroenterologist. The FMT is infused into the colon by performing a colonoscopy. FMT will be performed on Cycle 1 Day 1 and will take 15 to 30 minutes.
  Pembrolizumab, 200mg, through an IV over 30 minutes on Cycle 1 Day 1 (same day as the FMT), and then again on Day 1 of each 21-day cycle for an additional 3 cycles (Cycles 2 - 4).
  Interventions: Drug: Fecal Microbiota Transplant with Pembrolizumab

INTERVENTIONS:
Drug: Fecal Microbiota Transplant with Pembrolizumab — FMT is a procedure in which fecal matter or stool is collected from a tested donor, mixed with a saline or other solution, strained and infused into the colon by doing a colonoscopy. The FMT consists of introducing normal bacterial flora contained in stool collected from a donor into your small intestine. In this case, the donor is patient with advanced melanoma who has been treated with a PD-1 inhibitor (nivolumab or pembrolizumab) and has been rendered disease-free as a result. The FMT will be performed on Cycle 1 Day 1.
  Pembrolizumab, 200mg, through an IV over 30 minutes on Cycle 1 Day 1 (same day as the FMT, and then again on Day 1 of each 21-day cycle for an additional 3 cycles (Cycles 2 - 4).

SUMMARY:
The main goal of this research study is to determine if the fecal microbiota transplant (FMT) improves the body's ability to fight your cancer.

DETAILED DESCRIPTION:
This is a phase II Simon two-stage single-center study of concurrent fecal microbiota transplang (FMT) with pembrolizumab in patients with PD-1 resistant/refractory melanoma. The study will be conducted over a 12-week period (and up to 24-weeks in responding patients).

Patient eligibility is based upon prior exposure to PD-1 inhibitor therapy and response at first (or subsequent) restaging scans from week 12 up to week 52. Patients must have received a minimum of 2 cycles to be considered eligible. Patients who have received either nivolumab or pembrolizumab are eligible. Patients who have received pembrolizumab/nivolumab in combination with other investigational agent(s) may be eligible at the discretion of the treating investigator. PD-1 refractory disease is defined as progressive disease (PD) at the first (or subsequent) radiographic evaluation while receiving PD-1 inhibitor treatment as assessed by RECIST v1.1 on a restaging scan. Other eligibility criteria include absence of CNS disease, presence of disease amenable to biopsy and lack of contra-indications to FMT administration. Patients will be stratified on the presence or absence of liver metastases.

Suitable patients will be identified following first (or subsequent) restaging study that documents progressive disease (RECIST v1.1). Patients will undergo a screening evaluation consisting of imaging (including CNS if clinically suspected), tumor biopsy, and serological/stool studies to confirm suitability for FMT administration. Eligible patients will receive FMT endoscopically (along with intestinal biopsy) (with cycle 1 pembrolizumab +/- 3 days) followed by 3 further cycles of pembrolizumab (cycles 2-4) following which restaging will be performed. Patients with stable and/or responding disease will continue to receive pembrolizumab on study for 4 cycles. Patients with stable and/or responding disease after 8 cycles of pembrolizumab will continue to receive therapy off study until disease progression or up to two years from FMT administration.

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically or cytologically confirmed diagnosis of unresectable stage III or IV melanoma. Patient may not have a diagnosis of uveal or mucosal melanoma.
* Have received any number of prior systemic therapies for metastatic disease. Prior radiation therapy (any number) and interferon use (any formulation and/or duration) in the adjuvant or metastatic disease settings is permitted. Vaccine therapy will be counted as systemic therapy.
* Patient must currently be receiving systemic PD-1 immunotherapy with pembrolizumab or nivolumab to be eligible. Patients who have received PD-1 immunotherapy in the adjuvant setting and then replaced are eligible.
* Must be PD-1 inhibitor refractory/resistant - defined as having received at least 2 doses of pembrolizumab with documented systemic disease progression on staging imaging. PD will be defined as increase in tumor burden > 20% relative to nadir (minimum recorded tumor burden) by RECIST v1.1. Once PD is confirmed, initial date of PD documentation will be considered as the date of disease progression. Patients can be enrolled at any time following initiation of PD-1 therapy assuming they have not had (at any time) a record of response to PD-1 therapy (prior best response of stable disease - acceptable; prior best response of complete/partial response - unacceptable). For patients receiving adjuvant PD-1 inhibitor therapy, initial date of PD documentation will be considered as the date of disease progression.
* Patients with CNS progression (parenchymal but not leptomeningeal) are eligible if CNS metastases are treated and deemed stable (with a repeat CT/MRI imaging study) prior to the enrollment date. If radiation is used to treat CNS parenchymal disease, a 2 week washout period will apply (counted from Day 1 treatment). Stability must be confirmed with a repeat CT/MRI imaging study performed as part of the screening evaluation (at least 2 weeks after radiation). Patients with new CNS metastases identified during screening are ineligible.
* Consent to receive FMT administered endoscopically (colonoscopically) and undergo necessary bowel preparation pre-procedure.
* Understand infectious risks associated with FMT administration. Although FMT infusate has been screened for bacteria, viruses, fungi and parasites there is a risk of transmission of known and unknown infectious organisms contained in the donor stool. Post-FMT bacteremia (e.g. E. coli), sepsis and fatal events may rarely occur.
* Understand non-infectious risks associated with FMT administration. Possible allergy and/or anaphylaxis to antigens in donor stool; theoretical risk of developing disease possibly related to donor gut microbiota including but not limited to: obesity, metabolic syndrome, cardiovascular disease, autoimmune conditions, allergic/atopic disorders, neurologic disorders, psychiatric conditions and malignancy.
* Understand risks associated with colonoscopy including risk of infection transmission, colonic perforation, aspiration pneumonia, and death.
* Understand that data regarding the long-term safety risk of FMT are lacking.
* Consent to participate in the correlative studies and should have available tumor tissue for tumor biopsies. Acceptable biopsies include surgical biopsy, core biopsy or punch/surgical tumor biopsies (of accessible lesions).
* Have measurable disease as per RECIST version 1.1. At least 1 of the tumor sites must be amenable to biopsy and this may not be the site of disease used to measure antitumor response.
* Be willing and able to provide written informed consent for the trial.
* Be 18 years of age or older on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function:

Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment) Serum creatinine OR Measured or calculateda creatinine clearance (GFR can also be used in place of creatinine or CrCl) - ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for patients with liver metastases Albumin >2.5 mg/dL International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

* Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential must be willing to use an adequate method of contraception. Contraception, for the course of the study through 120 days after the last dose of study medication. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
* Male patients of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

- Presence of absolute contra-indications to FMT administration: Toxic megacolon Severe dietary allergies (e.g. shellfish, nuts, seafood) Inflammatory bowel disease Anatomic contra-indications to colonoscopy

* Patients receiving PD-1 therapy whose disease is responding or stable (as defined by RECIST v1.1).
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Highly symptomatic patients (e.g., declining ECOG performance status; rapidly worsening symptoms; rapid progression of disease; progression of tumor at critical anatomical sites (e.g., spinal cord compression) requiring urgent alternative medical intervention) are not eligible.
* Expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (> 10 mg prednisone daily or equivalent) or any other form of immunosuppressive therapy prior to trial treatment. Patients receiving systemic steroids at physiologic doses are permitted to enroll assuming steroid dose is not above the acceptable threshold (> 10 mg prednisone daily or equivalent).
* Has a known history of a hematologic malignancy, primary brain tumor or sarcoma, or of another primary solid tumor, unless the patient has undergone potentially curative therapy with no evidence of that disease for five years. NOTE: The time requirement also does not apply to patients who underwent successful definitive resection of basal or squamous cell carcinoma of the skin, superficial bladder cancer, in situ cancers including cervical cancer, breast cancer, melanoma, or other in situ cancers.
* Active central nervous system (CNS) metastases and/or leptomeningeal involvement. Patients with treated brain metastases will be re-screened (MRI brain or CT head with IV contrast). Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by MRI/CT for at least two weeks prior to the first dose of study drug), have no evidence of new or enlarging brain metastases and are off systemic steroids (≤ 10 mg/day prednisone or equivalent) for at least one weeks prior to enrollment. Patients with leptomeningeal disease (leptomeningeal enhancement on MRI/CT imaging and/or positive CSF cytology) are not eligible to enroll. Patients with no history of CNS disease will not require a repeat MRI brain unless they have symptoms to suggest new brain metastases.
* Had a severe hypersensitivity reaction to treatment with pembrolizumab or any of its excipients.
* Has an active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents. Patients with vitiligo, type I diabetes, resolved childhood asthma/atopy are exceptions to this rule. Patients who require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Patients with hypothyroidism stable on hormone replacement are not excluded from the study.
* Has a history of (non-infectious) pneumonitis that was life-threatening and/or required invasive support (CTCAE grade 4 or greater) or current pneumonitis.
* Has serious concomitant illnesses, such as: cardiovascular disease (uncontrolled congestive heart failure, hypertension, cardiac ischemia, myocardial infarction, and severe cardiac arrhythmia), bleeding disorders, autoimmune diseases, severe obstructive or restrictive pulmonary diseases, active systemic infections, and inflammatory bowel disorders. This includes HIV or AIDS-related illness, or active HBV and HCV.
* Has an active infection requiring systemic therapy.
* Has active COVID-19 infection and/or exposure to SARS-CoV-2 defined as Positive SARS-CoV-2 result on nasopharyngeal and/or stool specimens (by RT-PCR test), Active COVID-19 infection (per CDC guidelines), Exposure to active COVID-19 infected patient (as confirmed using SARS-CoV-2 RT-PCR test or other approved test) as defined per CDC guidelines
* Has active human immunodeficiency virus (HIV) infection (as manifested by presence of HIV 1/2 antibodies and/or positive HIV ELISA/Western Blot assays).
* Has active Hepatitis B or Hepatitis C infection. Patients with a history of Hepatitis B/C infection who have received anti-viral therapy and are disease free (Hep B - negative HBsAg and HBV DNA; Hep C - negative HCV RNA) may be considered for enrollment after discussion with Principal Investigator.
* Has a known history of active TB (Bacillus Tuberculosis).
* Patient has received a live vaccine within 4 weeks prior to the first dose of treatment.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

* Has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Patients with prior adverse events on replacement therapy who are asymptomatic or minimally symptomatic are not excluded from the study (i.e. hypothyroidism, hypopituitarism, adrenal insufficiency).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, Principal Investigator — Univ of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davar D, Dzutsev AK, McCulloch JA, Rodrigues RR, Chauvin JM, Morrison RM, Deblasio RN, Menna C, Ding Q, Pagliano O, Zidi B, Zhang S, Badger JH, Vetizou M, Cole AM, Fernandes MR, Prescott S, Costa RGF, Balaji AK, Morgun A, Vujkovic-Cvijin I, Wang H, Borhani AA, Schwartz MB, Dubner HM, Ernst SJ, Rose A, Najjar YG, Belkaid Y, Kirkwood JM, Trinchieri G, Zarour HM. Fecal microbiota transplant overcomes resistance to anti-PD-1 therapy in melanoma patients. Science. 2021 Feb 5;371(6529):595-602. doi: 10.1126/science.abf3363. PMID 33542131
- [Derived] Villemin C, Six A, Neville BA, Lawley TD, Robinson MJ, Bakdash G. The heightened importance of the microbiome in cancer immunotherapy. Trends Immunol. 2023 Jan;44(1):44-59. doi: 10.1016/j.it.2022.11.002. Epub 2022 Dec 1. PMID 36464584

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Microbiota Transplant (FMT) With Pembrolizumab: The FMT along with an intestinal biopsy will be performed as outpatient by a gastroenterologist. The FMT is infused into the colon by performing a colonoscopy. FMT will be performed on Cycle 1 Day 1 and will take 15 to 30 minutes.
  Pembrolizumab, 200mg, through an IV over 30 minutes on Cycle 1 Day 1 (same day as the FMT), and then again on Day 1 of each 21-day cycle for an additional 3 cycles (Cycles 2 - 4).
  Fecal Microbiota Transplant with Pembrolizumab: FMT is a procedure in which fecal matter or stool is collected from a tested donor, mixed with a saline or other solution, strained and infused into the colon by doing a colonoscopy. The FMT consists of introducing normal bacterial flora contained in stool collected from a donor into your small intestine. In this case, the donor is patient with advanced melanoma who has been treated with a PD-1 inhibitor (nivolumab or pembrolizumab) and has been rendered disease-free as a result. The FMT will be performed on Cycle 1 Day 1.
  Pembrolizumab, 200mg, through an IV over 30 minutes on Cycle 1 Day 1 (same day as the FMT, and then again on Day 1 of each 21-day cycle for an additional 3 cycles (Cycles 2 - 4).
Period: Overall Study
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the FMT recipient study
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.85 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Number of patients with patients with objective responses (Complete Response (CR) + Partial Response (PR), per RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 3 years
Population: All treated patients who were evaluable for radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 13
Participants
  Partial Response | 2
  Progressive Disease | 1

2. Secondary Outcome: Disease Control Rate (DCR)
Description: Number of patients with patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) per RECIST 1.1. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 3 years
Population: All treated patients who were evaluable for radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 13
Participants
  Partial Response (PR) | 2
  Stable Disease (SD) | 10
  Complete Response (CR) | 1

3. Secondary Outcome: Incidence of Grade III/IV Toxicities
Description: Number of patients who experienced grade III or grade IV toxicities per CTCAE v5.0, related to study treatment.
Time Frame: Up to 4 years
Population: All treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 2
Participants
  Atrial fibrillation | 1
  Lymphocyte count decreased | 1
  Arthralgia | 1
  Myopathy | 1
  Hyponatremia | 2

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from first response to to treatment until documented disease progression by RECIST v1.1 or death due to any cause. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Progressive Disease (PD): Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 4 years
Population: All treated patients who were evaluable for radiologic response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 11
months | 9 [3 to 32]

5. Secondary Outcome: 6-month Progression-free Survival (PFS)
Description: Percentage of patients who did not experience documented disease progression by RECIST v1.1 or death due to any cause from start of treatment until 6 months post treatment initiation. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 6 months
Population: All treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 10
percentage of participants | 61 [35 to 79]

6. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: Percentage of patients who did not experience documented disease progression by RECIST v1.1 or death due to any cause from start of treatment until 12 months post treatment initiation. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 12 months
Population: All treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 5
percentage of participants | 34 [13 to 57]

7. Secondary Outcome: 24-month Progression-free Survival (PFS)
Description: Percentage of patients who did not experience documented disease progression by RECIST v1.1 or death due to any cause from start of treatment until 24 months post treatment initiation. Progression as defined by RECIST v1.1 for target lesions: Progressive Disease (PD): smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). For non-target lesions: Appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: At 24 months
Population: All treated patients who were evaluable for radiologic response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 4
percentage of participants | 34 [13 to 57]

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS), defined as time from first dose of study treatment until death due to any cause.
Time Frame: Up to 6.5 years
Population: All enrolled patients followed for survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 20
months | 34 [6 to NA] — Upper bound of 95%CI not reached

9. Secondary Outcome: 6-month Overall Survival (OS)
Description: Percentage of patients alive at 6 months from first dose of study treatment.
Time Frame: At 6 months
Population: All study patients followed for survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 14
percentage of participants | 75 [49 to 89]

10. Secondary Outcome: 12-month Overall Survival (OS)
Description: Percentage of patients alive at 12 months from first dose of study treatment.
Time Frame: At 12 months
Population: All enrolled patients followed for survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 11
percentage of participants | 64 [39 to 81]

11. Secondary Outcome: 24-month Overall Survival (OS)
Description: Percentage of patients alive at 24 months from first dose of study treatment.
Time Frame: At 24 months
Population: All enrolled patients followed for survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
Number analyzed (Participants) | 10
percentage of participants | 64 [39 to 81]

12. Secondary Outcome: Change in T-cells Composition
Description: Quantitative differences in CD8 + PD1+ T cells (measured by percent of total cells) and MFI (staining intensity) between pre- and post- treatment samples from patients that respond and patients that do not respond (per RECIST 1.1), to study treatment.
  Information available in linked citation.
Time Frame: 4 years
Reporting Status: Not Posted

13. Secondary Outcome: Change in Innate/Adaptive Immune System Subsets
Description: Changes in CD8+ T-cell receptor diversity (quantified/determined by using Immunoseq analyses), CD4 + Foxp3 + T regulatory cells, CD56 + NK cells, CD68+ dendritic cells between pre- and post- treatment samples from patients that respond and patients that do not respond (per RECIST 1.1), to study treatment.
  Information available in linked citation.
Time Frame: 4 years
Reporting Status: Not Posted

14. Secondary Outcome: Function of T-cells
Description: Functional analyses (measured by percent of total cells) expressing IFNgamma) and MFI (staining intensity) between pre- and post- treatment samples from patients that respond and patients that do not respond (per RECIST 1.1), to study treatment.
  Information available in linked citation.
Time Frame: 4 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Association of PD-1 Response With (Common) Gut Microbiota
Description: Changes in bacterial abundance (quantified by the operational taxonomic unit (OTU)) which indicates the number of different species present along with the representative proportion of each species in the sample) and bacterial diversity (quantified by alpha diversity which is defined by the Shannon Index and quantifies both the organismal richness of a sample and the evenness of the organisms' abundance distribution), between pre- and post- treatment samples from patients that respond and patients that do not respond (per RECIST 1.1) to study treatment.
  Information available in linked citation.
Time Frame: 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: up to 6.5 years Serious and Adverse Events: up to 4 years
Arm/Group | Fecal Microbiota Transplant (FMT) With Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 14/20
Serious Adverse Events (participants affected / at risk) | 12/20
Other Adverse Events (participants affected / at risk) | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fecal Microbiota Transplant (FMT) With Pembrolizumab (N=20)
Acute kidney injury (Renal and urinary disorders) | 1/6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/6
Atrial fibrillation (Cardiac disorders) | 1/6
Depression (Psychiatric disorders) | 1/6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/6
Fall (Injury, poisoning and procedural complications) | 1/6
Failure to Thrive (General disorders) | 1/6
Hypercalcemia (Metabolism and nutrition disorders) | 1/6
Cellulitis (Investigations) | 1/6
specifymyopathy (Investigations) | 1/6
Localized edema (General disorders) | 1/6
Myopathy (Musculoskeletal and connective tissue disorders) | 1/6
Pain (General disorders) | 1/6
Peripheral motor neuropathy (Nervous system disorders) | 1/6
Rectal hemorrhage (Gastrointestinal disorders) | 1/6
Groin Abscess (Skin and subcutaneous tissue disorders) | 1/6
left hip closed reduction possible open reduction/revision (Surgical and medical procedures) | 1/6
left lateral hip excision (Surgical and medical procedures) | 1/6
resection of tumor (Surgical and medical procedures) | 1/6
right neck dissection (Surgical and medical procedures) | 1/6
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fecal Microbiota Transplant (FMT) With Pembrolizumab (N=20)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 6
Anemia (Blood and lymphatic system disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
B12 deficiency (Investigations) | 1
Bloating (Gastrointestinal disorders) | 1
bradycardia (Cardiac disorders) | 3
Constipation (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine increased (Investigations) | 3
creatinine increased (Investigations) | 1
decreased albumin (Investigations) | 1
decreased chloride (Investigations) | 1
Decreased protein (Investigations) | 1
decreased protein (Investigations) | 2
Decreased temperature (Investigations) | 1
decreased testosterone (Endocrine disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Delayed Wound Healing of biopsy site (Surgical and medical procedures) | 1
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 7
Dizziness (Nervous system disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
elevated TSH (Investigations) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2
Eye swelling (Eye disorders) | 1
Fall (Injury, poisoning and procedural complications) | 3
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Groin Abscess (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hemoptysis (Investigations) | 1
Hip Pain (General disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 2
hyperphosphatemia (Investigations) | 1
Hypertension (Vascular disorders) | 12
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 12
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hypovolemia (Investigations) | 1
ib fractures (Injury, poisoning and procedural complications) | 1
Inceased phos (Investigations) | 1
Increased Absolute Neutrophils (Investigations) | 1
increased bilirubin (Investigations) | 1
increased BUN (Investigations) | 3
increased creatinine (Metabolism and nutrition disorders) | 1
Increased LDH (Investigations) | 7
increased LDH (Investigations) | 5
increased phosphorus (Investigations) | 1
Increased Platelets (Investigations) | 1
Increased ptt (Investigations) | 1
Increased TSH (Investigations) | 2
increased TSH (Investigations) | 1
increased uric acid (Metabolism and nutrition disorders) | 1
Increased WBC (Investigations) | 1
Increased White blood cells (Investigations) | 1
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
intermittent weakness (Investigations) | 1
Knee pain (Investigations) | 1
LDH Increased (Investigations) | 2
LDH increased (Investigations) | 1
Leukocytosis (Investigations) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
Lung infection (Infections and infestations) | 3
Lymphocyte count decreased (Investigations) | 7
Lymphocyte count increased (Investigations) | 1
moonface (Investigations) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Myopathies (Musculoskeletal and connective tissue disorders) | 1
myopathy (Investigations) | 1
Nausea (Gastrointestinal disorders) | 5
Neutrophil count decreased (Investigations) | 4
Pain (General disorders) | 7
pain - bicep (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
pruritic mass - right lower flank (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Sinus bradycardia (Cardiac disorders) | 3
Sinus tachycardia (Cardiac disorders) | 1
Spinal Stenosis (Investigations) | 1
T6-T10 Spinal Infarct (Investigations) | 1
tachycardia (Cardiac disorders) | 2
Tremor (Nervous system disorders) | 2
troponin T increased (Investigations) | 1
TSH increased (Investigations) | 2
Tumor Lysis Syndrome (General disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vitiligo (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 3
Wound infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT03341143/Prot_SAP_000.pdf